CLINICAL TRIAL: NCT01943370
Title: Early Saline Irrigation to Decrease Post-operative Endoscopic Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Caroline Xu, Resident, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: ESESS-001; Pro00042764 (Other: HREB)
Record Dates: First submitted 2013-09-06; First posted 2013-09-17 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Rhinosinusitis
Keywords: endoscopic sinus surgery; post-operative irrigation; pain; debridement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early saline irrigation (Experimental): Initiation of early saline irrigation
  Interventions: Other: Early saline irrigation
- Late or Routine Saline Irrigation (Active Comparator): Routine initiation of saline irrigation
  Interventions: Other: Early saline irrigation; Other: Routine Irrigation

INTERVENTIONS:
Other: Early saline irrigation — Initiation of post-operative saline irrigation earlier during the post-operative course
Other: Routine Irrigation — Routine initiation of saline irrigation
  Arms: Late or Routine Saline Irrigation

SUMMARY:
Nasal saline is a common treatment adjunct in the post-operative setting for endoscopic sinus surgery. However, the ideal timing and quantity of irrigation in the early post-operative period remains unknown. Proposed benefits of early, large volume irrigation include removal and softening of crusts, resulting in improved mucociliary clearance. The potential benefit of early large volume saline irrigation on post-operative day three to ease or reduce the need for early post-operative debridement has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosis of CRS with or without polyposis
* Undergoing bilateral endoscopic sinus surgery
* Availability of pre-operative CT paranasal sinuses

Exclusion Criteria:

Patients with diagnosis of:

* Primary ciliary dyskinesia
* Immunodeficiency
* Cystic fibrosis

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pain | Early post-operative (Day 10)
  Pain and discomfort during early post-operative debridement on post-operative day 10

SECONDARY OUTCOMES:
Endoscopic appearance | Early (post-operative day 10)
  Early post-operative POSE score on post-operative day 10
Late endoscopic appearance at 6 months | 6 months
  Late post-operative endoscopic POSE score at 6 months